CLINICAL TRIAL: NCT05928988
Title: A Phase 1, Open-label, Fixed-sequence Study to Estimate the Effects of Multiple-dose Administration of Itraconazole on the Pharmacokinetics of SHR8554 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Itraconazole on Pharmacokinetics (PK) of SHR8554 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR8554-103
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR8554 and itraconazole (Experimental): SHR8554 will be provided in a solution. Participants will receive 1 mg SHR8554 by intravenous pump on Day 1 and Day 9.
  Itraconazole capsules 200 mg orally after meals twice daily for 7 days from Day 4 to Day 10.
  Interventions: Drug: SHR8554；Itraconazole

INTERVENTIONS:
Drug: SHR8554；Itraconazole — Drug: SHR8554 Administered as specified in the treatment arm Drug: Itraconazole Administered as specified in the treatment arm

SUMMARY:
This drug-drug interaction (DDI) study has been designed to characterize the pharmacokinetic profile of SHR8554 when co administered with a strong cytochrome P450 3A4 (CYP3A4) inhibitor itraconazole

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, aged 18 to 45 years (inclusive).
2. Female subjects body weight≥45 kg, male subjects body weight≥50 kg, body mass index (BMI) of 19.0 to 26.0 kg/m2 (inclusive).
3. Understand the study procedures in the informed consent form and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subjects with a history of drug allergy, or a history of specific allergies, or known allergy to SHR8554 or itraconazole or similar.
2. Any condition or disease detected during the medical interview/physical examination that would render the participant unsuitable for the study as determined by the investigator.
3. Subjects with positive tests for infectious diseases.
4. Subjects who have undergone major surgery within 3 months prior to screening or have undergone surgery that could significantly affect the in vivo course or safety evaluation of the study drug.
5. History of using any medication within 2 weeks prior to the first dosing.
6. Subjects who have received vaccination within 1 month prior to screening or plan to receive vaccination during the trial.
7. Excessive daily consumption of tea, coffee, grapefruit/grapefruit juice and other special diets in the 1 month prior to screening.
8. Subjects with a history of substance abuse, drug use or a positive screening test for substance abuse.
9. Female who are pregnant or breastfeeding, or have a positive pregnancy test.
10. Subjects who may not be able to complete the study for other reasons or who the investigator believes should not be included.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Cmax：observed maximum plasma concentration | Day 1 and Day 9 (pre-dose up to 48 hours post-dose)
AUC0-t ：area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration | Day 1 and Day 9 (pre-dose up to 48 hours post-dose)
AUC0-∞：area under the plasma concentration-time curve from time 0 to infinity | Day 1 and Day 9 (pre-dose up to 48 hours post-dose)
Tmax：observed time to reach Cmax | Day 1 and Day 9 (pre-dose up to 48 hours post-dose)
Vz ：apparent volume of distribution | Day 1 and Day 9 (pre-dose up to 48 hours post-dose)
MRT0-∞：mean residence time from time 0 to infinity | Day 1 and Day 9 (pre-dose up to 48 hours post-dose)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Baseline up to Day 18
Incidence of participants with clinical laboratory abnormalities | Baseline up to Day 18
Incidence of participants with vital signs abnormalities | Baseline up to Day 18
Incidence of participants with physical exam abnormalities | Baseline up to Day 18

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang L, Jiang H, Huang Y, Li J. Exploring Pharmacokinetic interactions between SHR8554, a micro-opioid receptor biased agonist, and Itraconazole in healthy Chinese subjects. Sci Rep. 2025 Jul 2;15(1):22635. doi: 10.1038/s41598-025-98697-3. PMID 40593123